CLINICAL TRIAL: NCT02444923
Title: A Randomised Controlled Research to Asses the Clinical Performance and Effect on Vision Related Quality of Life of Rigid Gas Permeable Scleral Versus Corneal Contact Lenses for Keratoconus and Other Irregular Cornea Disorders
Brief Title: Scleral Versus Corneal RGP Contact Lenses in Irregular Cornea Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London South Bank University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Levita
Record Dates: First submitted 2015-04-21; First posted 2015-05-15 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Irregular; Contour of Cornea; Keratoconus; Pellucid Marginal Corneal Degeneration; Injury of Cornea; Irregular Astigmatism
Keywords: Corneal rigid gas permeable contact lenses; Scleral rigid gas permeable contact lenses; Custom Scleral contact lenses; Keratoconus; Irregular cornea; Pellucid marginal degeneration; Post keratoplasty irregular cornea; Post refractive surgery irregular cornea; Traumatic irregular cornea
MeSH Terms: conditions — Keratoconus; Corneal Injuries

STUDY DESIGN:
Intervention Model Description: Randomised control trial with a 2x2 crossover
Who Masked: Investigator
Masking Description: The practitioner who measures the visual outcomes is naive to the type of lens the participant is wearing
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scleral rigid gas permeable contact lenses (Experimental): The experimental intervention is the Scleral Rigid Gas Permeable contact lens (SRGPcl), Zenlens™. These lenses are designed to bridge the cornea and fit in alignment with the sclera, thus avoiding any detrimental effects associated with corneal contact.
  Interventions: Device: Scleral rigid gas permeable contact lenses (SRGPcl) (Zenlens™); Device: Corneal Rigid gas Permeable contact lenses (CRGPcl) (Rose K2)
- Corneal rigid gas permeable contact lenses (Placebo Comparator): The control intervention is the RoseK2™ Corneal Rigid Gas Permeable contact lens (CRGPcl). Corneal lenses are considered the gold standard in the management of the visual disability due to keratoconus and other related irregular cornea disorders.
  Interventions: Device: Scleral rigid gas permeable contact lenses (SRGPcl) (Zenlens™); Device: Corneal Rigid gas Permeable contact lenses (CRGPcl) (Rose K2)

INTERVENTIONS:
Device: Scleral rigid gas permeable contact lenses (SRGPcl) (Zenlens™) — Custom manufactured scleral rigid gas permeable contact lenses. These lenses are designed to fit the eye with high level of precision. The aim is to bridge the cornea and fit in alignment with the sclera, thus avoiding any detrimental effects associated with the corneal rigid gas permeable lenses.
  Other Names: Scleral lenses; Zenlens; Custom Scleral Contact Lenses; RGP Scleral Lenses
Device: Corneal Rigid gas Permeable contact lenses (CRGPcl) (Rose K2) — The Rose K2 lens is a widely used corneal gas permeable lens designed for keratoconus and other irregular cornea disorders
  Other Names: Rose K2 corneal gas permeable contact lenses

SUMMARY:
The most common causes for irregular cornea (IC) in hospital contact lens practice are Keratoconus (KC) and related cornea thinning disorders. These conditions cause mild to marked impairment of vision and cannot be effectively corrected by spectacles and soft contact lenses. The gold standard in the management of KC is Corneal Rigid Gas Permeable contact lenses (corneal lenses), which correct approximately 90% of the corneal irregularity.

Compared with a normal cornea, the cornea in KC is irregular and this results in a compromise to the fit of rigid corneal lenses. Specifically, they bear on the cornea and this, together with the vulnerability of the cornea in KC, are implicated in corneal scarring, and disease progression as well as a significantly reduced vision related quality of life (QoL) in KC compared with corneal lens wearers who have no KC.

In cases where the compromise fit of corneal lenses proves problematic, large diameter Scleral RGP contact lenses (scleral lenses) may be used as a problem solver. Unlike the smaller corneal lenses which bear on the cornea, the scleral lenses completely bridge over the cornea and bear on the sclera.

The aim of this research is to investigate the performance of scleral lenses in KC participants who habitually wear corneal lenses.

The research question: is there a measurable difference in the visual performance and visual quality of life in participants with Irregular cornea disorders like keratoconus and other related conditions, who habitually wear corneal lenses in comparison with scleral lenses.

DETAILED DESCRIPTION:
The cornea is the transparent, fixed focus lens at the front of the eye. The cornea's curvature should be regular for good vision. The most common causes of irregular cornea (IC) in hospital contact lens practice are Keratoconus (KC) and related cornea thinning disorders. These conditions cause mild to marked impairment of vision due to High Order optical Aberrations (HOA), which degrade the retinal image quality and cannot be effectively corrected by spectacles and soft contact lenses. The gold standard in the management of KC are Corneal Rigid Gas Permeable contact lenses (corneal lenses), which correct approximately 90% of the corneal irregularity.

The corneal lenses fit differently in patients with a normal cornea compared to KC where they bear on the cornea. This fitting characteristic and the vulnerability of the cornea in KC are implicated in corneal scarring and disease progression as well as a significantly reduced vision related quality of life (QoL) in KC compared with corneal lens wearers who have no KC.

In cases where corneal lenses are not well tolerated, cause corneal insult, reduced visual performance or poor physical fitting characteristic, the large diameter Scleral RGP contact lenses (scleral lenses) may be used as a problem solver. Unlike the smaller corneal lenses which bear on the cornea, the scleral lenses completely bridge over the cornea and bear on the sclera.

The aim of this research is to investigate the performance of scleral lenses in participants who habitually wear corneal lenses.

Methodology The proposed quantitative experimental methodology is a randomised controlled trial (RCT) with cross over. The experimental intervention is a scleral RGP contact lens fitted from a fitting set and manufactured to exact specifications to optimise its physical fitting characteristics and optical performance. The control intervention is conventional design Corneal Rigid Gas Permeable contact lenses (corneal lenses). These lenses are considered the gold standard in the management of the visual disability caused by keratoconus and other IC disorders (Robertson, Cavanagh 2011).

Main inclusion criteria; patients aged 18-69 with irregular cornea disorder like keratoconus who wear corneal lenses.

Exclusion criteria: Patients who are satisfied and have good vision and comfort with soft contact lenses or spectacles.

Procedure After the consent procedure all subjects will undergo a National Eye Institute Visual Function Quality NEI-VFQ assessment and baseline Best Corrected Visual Acuity (BCVA) and Contrast Sensitivity Function (CSF) will be recorded.

Detailed fitting of an alternative type of corneal lenses and scleral lenses using a state of the art design of corneal and scleral RGP lens designs, which have been widely used in many clinics world-wide for some years. Appropriate clinical guidelines and best practice will be followed for the fitting and use of contact lenses. The lead applicant is a contact lens specialist who is highly experienced in fitting corneal and scleral RGP contact lenses.

Once the fitting has been completed the final lenses will be checked on eye at collection and will be checked after three weeks post collection of the best fitting lens and for the final results of visual performance and quality of life after 8-12 weeks of daily lens wear.

After this check up there will be a washout period of at least one month, during which the participants will wear their original corneal lenses before the wearing of the other intervention is started.

The crossover to the other lens will be implemented after the washout period. During this phase checkups will be performed in an identical manner to the first phase.

Lens designs and fitting The participants will initially be fitted with corneal lenses and scleral lenses to achieve an optimal fit. Horizontal and vertical displacement as well as angular scleral lens rotation would be measured to establish best lens parameters. The corneal lenses will be the Rose K™ design which is widely used all over the world and manufactured by Menicon David Thomas contact lens laboratory. The scleral lenses will be the Zenlens™, which is amenable to a wide variety of customised adjustments for fit optimisation, manufactured by UCO Lavec BV laboratory in the Netherlands.

Randomisation The research coordinator, colleague optometrist Anthony Stanton will randomise and register the participants to treatment and control groups. The participants and the chief investigator will be masked to the type of lens supplied.

Outcome measures Visual quality Two key measures of visual function, monocular best-corrected visual acuity (BCVA) and contrast sensitivity function (CSF) will be assessed at the beginning and the end of the lens wearing period and will constitute the outcome measures of this RCT. Both BCVA and CSF testing will use a commercially available instrument the CSV 1000E, which standardises test conditions and has been used in several research studies.

Quality of life The National Eye Institute-Visual Function Questionnaire (NEI-VFQ) (Mangione 2000) is a vision-related quality of life instrument designed to assess patients' perception of visual function and quality of life. This instrument, which has been used by other researchers investigating keratoconus (Kymes et al., 2004, 2008), will be applied as a baseline in the beginning of the study and at the completion of the period of use of each intervention.

Statistical and Data analysis A sample size calculation has been carried out that is based, conservatively, on a parallel trial design using data from previous research (Marsack, Parker et al. 2007, Nejabat, Khalili et al. 2012, Davis, Schechtman et al. 2006). The sample size calculation using the (Armitage and Berry, 1987) formula gives a required sample size of 15 participants in each group. The plan is therefore to continue the study until at least 30 have completed the study, 15 starting with scleral lenses and 15 with corneal lenses.

Preliminary checks will be carried out to ensure that there are no carry-over effects from the first to the second treatment periods, as recommended in the literature (Haynes et al., 2006; Wellek & Blettner, 2012).

We think it unlikely that there will be cross-over effects because the washout period should prevent this. However, in the unlikely event that there are significant washout effects or if a large proportion of participants drop out before the second treatment period then the study will be treated as a non-crossover RCT and the data from the first period will be analysed in the usual way as recommended by Haynes et al. (2006). Our conservative sample size calculation allows for this possibility.

If there is a satisfactory outcome to the preliminary checks then the study will be analysed as a cross-over RCT (Haynes et al., 2006; Wellek & Blettner, 2012).

Plan and timescale The length of participation in the study for each subject is anticipated not to exceed 5-7months during which time they are likely to be required to attend on 4-6 occasions. Study total length is anticipated to be from early 2015 to late 2016. The RCT will be conducted at the Central Middlesex Hospital (CMH) Ophthalmology Department where the lead researcher is a senior contact lens specialist optometrist.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of keratoconus or related corneal irregularity
* Age 18 years to 69 years.

Exclusion Criteria:

* Good visual quality with soft contact lenses and or spectacles

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10-25 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Monocular Best Corrected Visual Acuity (BCVA) | Baseline and after a minimum of 6 weeks of wear of each contact lens type, report at study completion
  High contrast BCVA will be measured by the specially constructed crowded, Logarithmic Minimum Angle of Resolution (LogMAR), Early Treatment Diabetic Retinopathy Survey (ETDRS) letter charts. An average score of 3 different, randomly presented charts will be taken as the final acuity score. It will be performed utilising the CSV1000E, under the established recommended standardised testing conditions utilised in a multitude of research protocols.

SECONDARY OUTCOMES:
Contrast Sensitivity Function | Measure at recruitment (Baseline), subsequent measurement after 6 weeks of wear, of lens 1 and 6 weeks of wear of lens 2. Study completion after 6-12 months.
  The Contrast Sensitivity Function (CSF) will be assessed at each of the four spatial frequencies 3, 6, 12 and 18 Cycles Per Degree (CPD) averaging the results from 2 different charts with sinusoidal grating patterns. This will be performed utilising the CSV1000E, under the established recommended standardised testing conditions utilised in a multitude of research protocols.
The National Eye Institute-Visual Function Questionnaire (NEI-VFQ) | Measure at recruitment (Baseline), subsequent measurement after 6 weeks of wear, of lens 1 and 6 weeks of wear of lens 2. Study completion after 6-12 months.
  The National Eye Institute-Visual Function Questionnaire (NEI-VFQ) (Mangione 2000) is a vision-related quality of life instrument designed to assess patients' perception of visual function and quality of life. The measurements include general health, general vision, ocular pain, near and distance activities, driving, colour vision, and peripheral vision. There are four components of psychological well being, these are; social function, mental health, role difficulties, and dependency function. It has been used to characterize the quality of life for patients with uveitis, diabetic retinopathy, glaucoma, and age-related macular degeneration (Mangione, Lee et al. 2001)
The Levit Subjective Comfort and Vision Scales | Measure at recruitment (Baseline), subsequent measurement after 6 weeks of wear, of lens 1 and 6 weeks of wear of lens 2. Study completion after 6-12 months.
  The Levit Subjective Comfort Scale (LSCS) and The Levit Subjective Vision Scale (LSVS) are Likert like scales which grade the participants' perception of their comfort and vision in contact lenses, on a scale from 1( worse) to 10 (best).
The final lens choice | At study completion after 6-12 months
  Each participant chose one of the two experimental lenses they wished to keep for future habitual use

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Levit, FCOptom, Principal Investigator — London South Bank Unversity; Martin Benwell, PhD, Study Director — London South Bank University; Bruce Evans, PhD, Study Chair — Institute of Optometry
Locations (1):
- Central Middlesex Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Visser ES, Van der Linden BJ, Otten HM, Van der Lelij A, Visser R. Medical applications and outcomes of bitangential scleral lenses. Optom Vis Sci. 2013 Oct;90(10):1078-85. doi: 10.1097/OPX.0000000000000018. PMID 23974663
- See also: Institute of Optometry — http://www.ioo.org.uk